CLINICAL TRIAL: NCT03616366
Title: The Mechanism and Prognosis of Pulmonary Circulation Dysfunction in Pulmonary Injury and Recovery
Brief Title: The Mechanism and Prognosis of Pulmonary Circulation Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2017-I2M-1-009
Record Dates: First submitted 2018-01-04; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: VTE
Keywords: VTE; SNP; biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — serum and blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous thromboembolism (VTE) is a condition which influenced by both environmental and genetic factors. This study is going to explore new significant Single nucleotide polymorphisms (SNPs) associated with VTE by Genome-Wide Association Studies (GWAS) and bioinformatics analysis. Transcriptomics and cytokine antibody array are also used to find new biomarkers of VTE's early diagnosis, severity and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Han population older than 14 years old
* Acute VTE patients diagnosed in 1 month
* With informed consent

Exclusion Criteria:

* Patients with psychosis
* Patients with contraindications for computed tomographic pulmonary angiography (CTPA)
* Chronic VTE
* Recurrence of chronic VTE

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Acute VTE patients and healthy controls
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-10 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause death | 6 months
  death

SECONDARY OUTCOMES:
Venous thromboembolism (VTE) recurrence | 6months
  VTE recurrence detected by echocardiography or CTPA scan
chronic thromboembolism pulmonary hypertension(CTEPH) | 6 months
  newly developed CTEPH detected by pulmonary angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Institute and Fu Wai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided